CLINICAL TRIAL: NCT06850519
Title: A Study and Biobank to Identify Genetic Risk Factors in the Pathogenesis of the Sneddon Syndrome
Brief Title: Genetic Risk Factors of the Sneddon Syndrome
Status: Completed | Type: Observational
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: Medical University of Vienna (Other); Unidade Local de Saúde de Coimbra, EPE (Other); Instituto de Investigación Marqués de Valdecilla (Other); Technical University of Munich (Other); Alfried Krupp Krankenhaus (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 1016/2021
Record Dates: First submitted 2021-09-08; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2021-09

CONDITIONS: Sneddon Syndrome
MeSH Terms: conditions — Sneddon Syndrome | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Sneddon: Whole exome sequencing
  Interventions: Genetic: Exome Sequencing and Sanger Sequencing

INTERVENTIONS:
Genetic: Exome Sequencing and Sanger Sequencing — Exome Sequencing and Sanger Sequencing

SUMMARY:
Sneddon syndrome (SS) is a rare disorder with an incidence of about 4/million/year that affects mainly young and predominantly female adults. It is characterized by recurrent strokes and livedo reticularis, a purple reticular patterning of the skin. A genetic predisposition to this disease, for which there is still no single therapy, is being discussed. Our group recently identified a homozygous nonsense mutation within epidermal growth factor repeat (EGFr) 19 of NOTCH3 in two siblings of a consanguineous family with Sneddon syndrome and pediatric stroke. In an attempt to find other possible contributing genes in Sneddon syndrome patients with adult-onset stroke, we also searched for loss-of-function variants in genes downstream of NOTCH3. In doing so, we found 2 patients carrying heterozygous loss-of-function variants in the PALLD and ANGPTL4 genes. Our results suggest that a bi-allelic loss-of-function mutation in NOTCH3 is a cause of familial Sneddon syndrome with pediatric stroke and that impaired NOTCH3 signaling is an underlying disease mechanism in general. In addition, we have identified several other promising variants that are either located in genes associated with NOTCH3 signaling or play a role in vascular function and stroke.

Based on these results, we now want to investigate whether these aforementioned variants are detectable in a larger number of patients and additionally analyze whether other genetic variants also play a role in disease pathogenesis. The goal of our project is to identify risk variants for Sneddon syndrome by whole exome sequencing and subsequent conventional sequencing....

The detection of a risk gene would be a helpful tool for the diagnosis of Sneddon syndrome and a possible basis for new therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18years old.
* Affected subjects must have been clinically diagnosed with Sneddon Syndrome. When analyzing families with Sneddon syndrome, healthy family members and participants with only symptoms of the skin will be included if consent is obtained.Frau Elli Greisenegger
* Unaffected subjects or subjects with symptoms restricted to the skin must have at least one family member with the clinical diagnosis Sneddon syndrome participating in the study.
* Subjects must be able to communicate well with the investigator, to understand the requirements of the study, as well as to understand and sign thewritten informed consent(= informed consent approved by thelocalethics committee).

Exclusion Criteria:

- Subjects who are unable to communicate well with the investigator, to understand the requirements of the study, as well as to understand and sign the written informed consent, are not eligible for inclusion in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Sneddon syndrome based on standard diagnosis criteria of Sneddon syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
potential genetic risk factor for Sneddon Syndrome present | 18 months
  occurence of genetic variants in genes associated with Sneddon Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Karl Landsteiner University, Sankt Pölten, Austria

IPD SHARING:
Plan to Share IPD: No